CLINICAL TRIAL: NCT01943227
Title: Effect of Alveolar Minute Ventilation on Respiratory Gas Heat Content
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 483184
Record Dates: First submitted 2013-09-11; First posted 2013-09-16 (Estimated); Results first posted 2019-10-28 (Actual); Last update posted 2019-10-28 (Actual); Status verified 2019-10

CONDITIONS: Ventilation Perfusion Mismatch
Keywords: humidity; enthalpy; mechanical ventilation
MeSH Terms: interventions — Tidal Volume

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 6ml/kg: Enthalpy measured in patients receiving controlled positive pressure ventilation 6ml/kg Tidal volume.
  The VQm monitor samples the gas at a rate of 3 L/min, returning the analyzed gas to the circuit. As the exhaled gas passes through the analytical chamber, the temperature and humidity are measured essentially continuously (40Hz). These data are combined with pressure measurements to determine the exhaled gas volume and then the heat content (enthalpy) is calculated.
  Interventions: Other: controlled positive pressure ventilation 6ml/kg tidal volume
- 9ml/kg: Enthalpy measured in patients receiving controlled positive pressure ventilation 9ml/kg Tidal volume.
  The VQm monitor samples the gas at a rate of 3 L/min, returning the analyzed gas to the circuit. As the exhaled gas passes through the analytical chamber, the temperature and humidity are measured essentially continuously (40Hz). These data are combined with pressure measurements to determine the exhaled gas volume and then the heat content (enthalpy) is calculated.
  Interventions: Other: controlled positive pressure ventilation 9ml/kg tidal volume

INTERVENTIONS:
Other: controlled positive pressure ventilation 9ml/kg tidal volume — controlled positive pressure ventilation 9ml/kg tidal volume
  Groups: 9ml/kg
Other: controlled positive pressure ventilation 6ml/kg tidal volume — controlled positive pressure ventilation 6ml/kg tidal volume
  Groups: 6ml/kg

SUMMARY:
This is a single site, prospective, non-blinded, non-randomized, non-interventional study designed to evaluate the effect of changes in alveolar minute ventilation on the measurement of respiratory heat loss (enthalpy).

DETAILED DESCRIPTION:
This is a single site, prospective, non-blinded, non-randomized, noninterventional study designed to evaluate the effect of changes in alveolar minute ventilation on the measurement of respiratory heat loss (enthalpy). Each patient will serve as their own control. The study will enroll adult patients without cardiac or respiratory illness. It is designed to evaluate the effect of the ventilatory pattern (tidal volume, rate) on respiratory heat loss measured using the VQm™ monitor during standard intra-operative clinical care that requires positive pressure ventilation (PPV)

ELIGIBILITY:
Inclusion Criteria:

* age greater than 18 years
* scheduled for an elective surgical procedure with an anticipated duration of more than 2 hours requiring general anesthesia and positive pressure ventilation using an endotracheal tube
* patient status ASA 1, 2 or 3
* no significant cardio-vascular or respiratory disease
* supine surgical position

Exclusion Criteria:

* Adults unable to give primary consent
* age less than 18 years
* pregnancy
* prisoners
* pre-existing cardiac or pulmonary disease
* infusion of inotropic drugs
* positive end expiratory pressure (PEEP) requirements >8 cm H2O
* increased intra-abdominal pressure (e.g. planned surgical pneumoperitoneum or ascitis)
* intra-operative patient position other than supine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients without cardiac or respiratory illness
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2013-08; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neal Fleming, MD, PhD, Principal Investigator — Professor, Anesthesiology & Pain Medicine
Locations (1):
- UC Davis Health System, Sacramento, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient recruitment and informed consent will be obtained in the UCDMC perioperative suite. Recruitment will be by direct discussion between the prospective candidates and the study investigators prior to their scheduled surgical procedure. The investigators will provide the consent form in person and give subject time to discuss with family.
Pre-assignment Details: The screening of patients will require the investigators to access personal health information to identify prospective subjects without HIPAA authorization. The research could not be practicably carried out without this waiver of consent. The risk of harm from contacting the participants is greater than the risk of the study procedures.
Groups:
- Large Tidal Volume; Smal Tidal Volume: Change in airway heat content
Period: Overall Study
Arm/Group | Large Tidal Volume | Smal Tidal Volume
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The study will enroll adult patients without cardiac or respiratory illness.
Groups:
- Large Tidal Volume; Small Tidal Volume: Airway heat content
- Total: Total of all reporting groups
Arm/Group | Large Tidal Volume | Small Tidal Volume | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] — The study will enroll adult patients without cardiac or respiratory illness.
  Years | 44 (10.8) | 42 (13.8) | 43 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 9
  Male | 4 | 7 | 11
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Airway Enthalpy
Description: This is a single site, prospective, non-blinded, non-randomized, non-interventional study designed to evaluate the effect of changes in alveolar minute ventilation on the measurement of respiratory heat loss (enthalpy) in Joules per minute.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Joules/Minute
Arm/Group | Large Tidal Volume | Smal Tidal Volume
Number analyzed (Participants) | 10 | 10
Joules/Minute | 32 (9.1) | 23 (8.9)

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | Large Tidal Volume | Small Tidal Volume
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes